CLINICAL TRIAL: NCT03642457
Title: Comparison Between Serratus Plane Block And Local Surgical Infiltration In Robotic Video Assisted Thoracoscopic Surgery- A Randomised Controlled Trial
Brief Title: Efficacy Between Serratus Plane Block And Local Infiltration In Vats
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution and unable to find new PI
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Yan Lai, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-1294
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer
Keywords: Video assisted thoracoscopic surgery; Serratus plane block; local infiltration
MeSH Terms: conditions — Lung Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, surgeon, and anesthesiologist in the case will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Serratus Plane Group (Active Comparator): Patients randomized to the group will receive a total 20cc of solution consisting of 0.5% bupivacaine with 133mg of liposomal bupivacaine injected in the serratus plane with the help of an ultrasound.
  Interventions: Drug: Bupivacaine; Drug: Bupivacaine liposome
- Placebo Group (Placebo Comparator): Patients randomized to the group will receive a total 20cc of 133mg liposomal bupivacaine injected prior to skin closure at the incision site as per surgeon's practice.
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine — 20 cc 0.5%
  Arms: Serratus Plane Group
Drug: Bupivacaine liposome — 133mg liposomal bupivacaine

SUMMARY:
Robotic video-assisted thoracoscopic surgery (VATS) is increasingly being used as it is a less invasive surgery compared to traditional methods, but the acute pain at an early stage after VATS has a major impact on perioperative outcomes. Effective post operative analgesia is believed to reduce morbidity, quicken recovery, improve patient outcome and reduce hospital costs. The site and extent of the incision influences the degree of pain due to disruption of intercostal nerves as well as inflammation of chest wall and pleura. Neuraxial and systemic opioids have been a gold standard as a part of multimodal analgesia for thoracic surgeries. Numerous modalities have been studied: thoracic paravertebral nerve blocks, thoracic epidural analgesia, intercostal nerve blocks, patient controlled analgesia (PCA), cryo-analgesia, transcutaneous electrical nerve stimulation (TENS), inter-pleural blocks, stellate ganglion blocks, long thoracic nerve blocks, and infiltration under direct vision by the surgeon.

Serratus plane block is an emerging regional technique that has proven to be effective in comparison to paravertebral blocks in patients undergoing breast surgery and mastectomy with reduced perioperative opioid consumption and improved pain scores.

The lateral pectoral nerve, medial pectoral nerve, intercostal nerves and long thoracic nerve are all targets for the serratus plane block. It can be safely performed under ultrasound guidance.

The purpose of the study is to evaluate the difference in quality of analgesia between efficacy of serratus plane block and local surgical infiltration by surgeon as measured by patient opioid consumption and pain scores.

DETAILED DESCRIPTION:
Participants will be assigned randomly using a computer-generated table of numbers to either serratus group or infiltration group. Block team will perform all blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology) class I-IV
* age 81-75

Exclusion Criteria:

* ASA class V
* morbid obesity
* patient refusal
* patients with chronic pain or on pain medications
* allergy to LA
* patients receiving any additional regional techniques
* coagulopathy
* patients receiving systemic anticoagulation
* local infection
* procedures anticipated to last more than 5 hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lai, MD, MPH, Principal Investigator — cahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai St. Luke's Hospital, New York, New York
  - Mount Sinai West Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Thoracic paravertebral block versus pectoral nerve block for analgesia after breast surgery. Egypt J Anaesth. 2013; 30: 129-135. Wahba, SS and Kamal, SM.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Serratus Plane Group | Placebo Group
Started | 35 | 30
Completed | 35 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serratus Plane Group | Placebo Group | Total
Number analyzed (Participants) | 35 | 30 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.29 (17.24) | 64.30 (11.01) | 58.37 (15.60)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing data
  Participants
    number analyzed (Participants) | 35 | 29 | 64
    Female | 18 | 18 | 36
    Male | 17 | 11 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 0 | 10
  Black or African American | 10 | 10 | 20
  Hispanic or Latino | 5 | 10 | 15
  White | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Amount of Opioid Consumption
Description: The amount of opioid consumption (in mg IV morphine equivalents) postoperatively up to 24 hours after the procedure.
Time Frame: up to 24 hours post procedure
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 35 | 30
MME | 18.93 (19.16) | 13.21 (18.93)

2. Secondary Outcome: Time to First Dose of Narcotic Administration
Description: Time to first dose of narcotic administration post procedure
Time Frame: up to 24 hours post procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 35 | 30
hours | 2.86 (4.17) | 3.09 (3.85)

3. Secondary Outcome: PACU Length of Stay
Description: The length of stay post procedure in the PACU
Time Frame: average 3-4 hours post procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 35 | 30
hours | 3.45 (2.41) | 3.05 (1.66)

4. Secondary Outcome: ICU Length of Stay
Description: The length of stay post procedure in the or ICU
Time Frame: up to 40 hours post procedure
Population: only those participants who required an ICU stay
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 7 | 3
hours | 32.57 (28.32) | 40.00 (27.71)

5. Secondary Outcome: Visual Analogue Score (VAS)
Description: Visual Analogue Score (VAS) pain score from 0 (no pain) to 10 (most pain)
Time Frame: up to 24 hours post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 35 | 30
score on a scale
  baseline | 2.31 (3.56) | 2.80 (3.65)
  at 2 hours | 3.09 (2.85) | 3.07 (2.57)
  at 6 hours | 3.03 (2.71) | 3.23 (3.02)
  at 18 hours | 2.17 (2.94) | 2.17 (2.73)
  at 24 hours | 1.89 (2.26) | 1.93 (2.57)

6. Secondary Outcome: Patient Satisfaction Score
Description: Patient satisfaction score from 0 (not satisfied) to 10 (extremely satisfied)
Time Frame: up to 24 hours post procedure
Population: Data not collected
Arm/Group | Serratus Plane Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Serratus Plane Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/30
Other Adverse Events (participants affected / at risk) | 0/35 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03642457/Prot_SAP_000.pdf